CLINICAL TRIAL: NCT06362707
Title: A Placebo Controlled Randomized Double-blind Parallel Group 12-month Trial of Fasudil for the Treatment of Early Alzheimer's Disease (FEAD)
Brief Title: Fasudil Trial for Treatment of Early Alzheimer's Disease (FEAD)
Acronym: FEAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University of Exeter (Other); Helse Fonna (Other); St. Olavs Hospital (Other); University Hospital, Akershus (Other); Haraldsplass Deaconess Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2023161001
Record Dates: First submitted 2024-02-02; First posted 2024-04-12 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-04

CONDITIONS: Cognitive Decline, Mild; Alzheimer Disease
Keywords: Alzheimer Disease; Mild Cognitive Decline; Fasudil
MeSH Terms: conditions — Cognitive Dysfunction; Lymphoma, Follicular; Alzheimer Disease | interventions — fasudil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasudil (Experimental): In recognition that fasudil has only been evaluated in published studies for treatment durations of up to 3 months, we intend to enroll participants in three successive cohorts of 20, 50 and 130 people, respectively. Participants in the initial cohort will undergo a 2-week titration period (60 mg total daily dose; 20 mg tds) before being escalated to the maintenance dose (120 mg total daily dose; 40 mg tds) for up to 50 additional weeks of treatment. The selected dose of 120mg per day is optimized for potential efficacy over the planned 12-month treatment period, while providing a reasonable margin of safety based on available clinical and nonclinical data.
  Interventions: Drug: Fasudil
- Placebo (Placebo Comparator): Following screening procedures, subjects will be randomized at baseline to receive fasudil or matching placebo across all cohorts. 1:1 randomization will be performed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fasudil — A ROCK inhibitor approved for treating vasospasms following subarachnoidal bleeding in Japan and China. Dosage: Participants will undergo a 2-week titration period at 60 mg daily before escalating to a maintenance dose of 120 mg daily.
  Arms: Fasudil
Drug: Placebo — Placebo tablets that look identical to the fasudil tablets and will follow the same dosing schedule as participants receiving fasudil.
  Arms: Placebo

SUMMARY:
The goal of this placebo-controlled double-blind Phase 2 clinical trial is to test in people with early Alzheimer's Disease.

The main questions it aims to answer are:

* Does treatment with fasudil, a ROCK-inhibitor, lead to significant improvement in working memory (based on computer-based working memory composite scores) compared to placebo in individuals with early Alzheimer's disease (AD) over 12 months?
* What is the effect of fasudil treatment for 12 months on other cognitive functions, brain metabolism measured by Fluorodeoxyglucose Positron Emission Tomography (FDG-PET), and other relevant clinical functions and biomarkers in individuals with early Alzheimer's disease (AD)?
* Treatment will be escalated to a maintenance dose of 120 mg total daily dose for up to 50 weeks, with regular clinic visits for efficacy and safety evaluations.
* Assessments will include cognitive tests, FDG-PET scans, and biomarker analyses, with follow-up by the Data and Safety Monitoring Board for ongoing safety review.

The study will compare participants receiving fasudil with those receiving placebo to see if fasudil treatment leads to improvements in cognitive functions, brain metabolism measured by FDG-PET.

DETAILED DESCRIPTION:
This is a 2-arm, parallel-group, 12-month, randomized, placebo-controlled double-blind Phase 2 trial of fasudil in up to 200 people with early AD. Fasudil is a ROCK-inhibitor (rho-associated protein kinase inhibitor), a vasodilator that is approved for treating vasospasms following subarachnoidal bleeding in Japan and China. The drug has acceptable safety and tolerability and has been shown to protect neurons and synapses in animal models of AD. Eligible participants must have Stage 3-4 mild cognitive impairment (MCI) or mild dementia due to AD, as recently defined by FDA Guidance, and have shown a significant change on a validated AD biomarker (e.g. amyloid PET scans or CSF Aβ 1-42 or blood p-tau 217 levels). In addition, they must have a CDR Global rating of 0.5 or 1.0 and an MRI scan within the past two years that has no findings inconsistent with AD.

People who meet all inclusion criteria will be enrolled in three successive cohorts of 20, 50, and 130 people, respectively. Participants will be randomized 1:1 to receive fasudil or a matching placebo. All participants will undergo a 2-week titration period at a total daily dose of 60 mg (20 mg tds) before being escalated to the maintenance dose of 120 mg total daily dose (40 mg tds) for up to 50 additional weeks of treatment. The selected dose of 120 mg per day is optimized for potential efficacy over the planned 12-month treatment while providing a reasonable margin of safety based on available clinical and nonclinical data. Participants will visit the clinic for efficacy and/or safety evaluations at 2-week intervals for the first month and then monthly thereafter (see Table 1. Schedule of Assessments).

The Data and Safety Monitoring Board (DSMB) will perform an unblinded review of the safety and pharmacokinetic (PK) data once all ongoing patients in Cohort 1 have completed at least 3 months of treatment and make recommendations to the study team that may include stopping or continuing the study (with or without changes to the study procedures).

The DSMB will continue to review all data available from Cohorts 1-3 for the remainder of the study at 3-monthly intervals, or more frequently if warranted by emergent data, and recommend any changes to the study procedures to ensure appropriate safety oversight and management of study participants through completion of the study.

The primary efficacy outcome is the FLAME (Factors of Longitudinal Attention, Memory and Executive Function) computer-based working memory composite. The key secondary outcomes are based on the expression of the AD-like hypometabolic pattern on FDG-PET and additional cognitive tests from the FLAME battery, including memory, working memory, attention, and executive functions. Additional secondary outcomes include CSF and blood-based AD biomarkers, and clinical measures including Clinical Global Impression of Change (CGIC), and Clinical Dementia Rating (CDR), neuropsychiatric symptoms (NPI), instrumental activities of daily living (Amsterdam IADL scale) and quality of life (DEMQOL). Standard safety measures include monthly assessments of adverse events (AEs), vital signs, and laboratory tests (including blood and urine analyses) as well as ECGs and the Columbia-Suicide Severity Rating Scale (C-SSRS).

ELIGIBILITY:
Inclusion Criteria:

* Early AD, eg Stage 3 MCI or Stage 4 (mild AD dementia), as recently defined by the FDA (2018; Figure 2)
* A significant change on a validated AD amyloid or tau biomarker (as determined either by visual reading of amyloid PET scans using any of the approved ligands, or CSF Aβ 1-42 levels or blood p-tau 217 cut-offs as determined by the clinical research laboratory)
* A CDR Global rating of 0.5 or 1.0 (Morris 1993) and have an MRI scan within the past two years that has no findings inconsistent with AD
* Capacity to give informed consent based on the clinical judgement of an experienced clinician
* The participant needs to have a reliable study partner with regular contact (a combination of face-to-face visits and telephone contact is acceptable) who has sufficient interaction with the participant to provide meaningful input into rating scales
* Age from 50 years
* Fluency in Norwegian and evidence of adequate premorbid intellectual functioning
* Capable of participating in all scheduled evaluations and complete all required tests
* Female participants must be of non-childbearing potential or have a negative serum pregnancy test within 14 days of baseline assessments and agree to the use of effective birth control throughout their participation in the study

Exclusion Criteria:

* Significant cerebrovascular disease, as indicated by clinical history, neurological examination, or on MRI (including cortical infarction or deep white matter or periventricular white matter hyperintensities with a Fazekas scale score of 3 (Fazekas et al 1987).
* A history of cerebrovascular bleeding or severe bleeding of the digestive tract, lungs, nose or skin
* Severe renal impairment (GFR <30) or serum creatinine or urea nitrogen values ≥3 times Upper normal limit (ULN) at screening or baseline
* Moderate to severe hepatic impairment. Serum alanine transaminase (ALT) or aspartate transaminase levels ≥3 times ULN at screening or baseline
* Currently poorly controlled diabetes as indicated by HbA1c values >9
* White blood cell (WBC) values <3.5 K/μl
* History of paralytic ileus or current severe chronic constipation
* Known allergy to fasudil or established systemic inflammatory disease or autoimmune disease.
* Clinically significant hypotension defined by blood pressure values <90/60 mmHg, regardless of the individual's sitting or standing position and associated with relevant clinical symptoms (e.g., tachycardia, dizziness, syncope)
* Current clinically significant depression or other mental disorder likely to affect cognition or interfere with study participation
* Recent (within 3 months) relevant medication changes. Participants must have been on stable anti-dementia (cholinesterase inhibitors or memantine) or anti-depressive medications for at least three months before the study
* Participants using sedating drugs, if unavoidable, will be excluded from the study. However, short-acting sleep medications can be used if taken as recommended and if the participant has maintained stability on them for a minimum of 3 months prior to the start of the study
* Participation in other drug trials
* Currently ongoing life-threatening disease, such as metastatic cancer, advanced cardiovascular disease, advanced respiratory disease, terminal kidney disease, or advanced stages of infectious diseases
* Any current or past neurological disease unrelated to Alzheimer's disease with cognitive sequelae
* A Corrected QT (QTc) interval ≥ 460 milliseconds for males or ≥ 470 milliseconds for females will be considered abnormal during the ECG assessments

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Cognition | The cognitive battery will be performed at baseline and every three months until last visit, supported by trial staff (up to 1 year).
  The primary outcome will be the FLAME computer-based working memory composite comprised of tests of working memory and episodic memory
Brain metabolism | The outcome will be change in FDG-PET between baseline and at 12 months.
  FDG-PET is a highly sensitive means of determining brain metabolism and has been accepted as a good proxy measure of synaptic function. Importantly, FDG-PET based measures of brain metabolism correlate well with cognitive decline in AD, better than amyloid plaques. Data from the Alzheimer's Disease Neuroimaging Initiative (ADNI) study suggest that FDG PET has good power to detect a 25% treatment effect over 12 months

SECONDARY OUTCOMES:
Plasma levels of ptau217 | Collection of blood samples will occur at baseline and the 12-month visit.
  This study involves the collection of blood samples, following standardized procedures. Blood markers associated with Alzheimer's disease (AD) will be analyzed for typical AD features to fulfill inclusion criteria. The primary focus will be on examining changes in levels of plasma ptau217 and nfl, measured in pg/mL.
Plasma levels of nfl | Collection of blood samples will occur at baseline and the 12-month visit.
  This study involves the collection of blood samples, following standardized procedures. Blood markers associated with Alzheimer's disease (AD) will be analyzed for typical AD features to fulfill inclusion criteria. The primary focus will be on examining changes in levels of plasma ptau217 and nfl, measured in pg/mL.
Levels of cerebrospinal Aβ1-40 and Aβ1-42 | Collection of CSF samples will occur at baseline and the 12-month visit.
  This study involves the collection of cerebrospinal fluid (CSF) samples, following standardized procedures. CSF markers associated with Alzheimer's disease (AD) will be analyzed for typical AD features, measured in pg/mL.
Levels of cerebrospinal tau and p-tau | Collection of CSF samples will occur at baseline and the 12-month visit.
  This study involves the collection of cerebrospinal fluid (CSF) samples, following standardized procedures. CSF markers associated with Alzheimer's disease (AD) will be analyzed for typical AD features, measured in pg/mL.
Blood pressure (Safety assessments) | Conducted at all visits throughout the 12-month duration of the study. Additionally, the Columbia Suicide Severity Rating Scale (C-SSRS) will be administered at screening, month 6, and month 12
  Safety measurements, blood pressure measured in millimetres of mercury (mmHg).
Pulse (Safety assessments) | Conducted at all visits throughout the 12-month duration of the study.
  Safety measurements, including pulse frequency in beats per minute (bpm).
Urine testing (Safety assessments) | Conducted at baseline and all visits throughout the 12-month duration of the study.
  Urine will be tested with a dipstick test to explore proteinuria or hematuria.
Blood urea nitrogen (BUN) (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in mmol/L
Potassium (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in mmol/L
Sodium (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in mmol/L
Calcium (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in mmol/L
Glucose (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in mmol/L
Hemoglobin (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in g/dL
Creatinine (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in μmol/L
Total and direct bilirubin (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in μmol/L
CRP (C-reactive protein) (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in mg/L
Aspartate aminotransferase (AST) (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in U/L (units per liter)
Serum glutamic-oxaloacetic transaminase (SGOT) (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in U/L (units per liter)
Alanine aminotransferase (ALT) (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in U/L (units per liter)
Serum glutamic-pyruvic transaminase (SGPT) (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in U/L (units per liter)
Alkaline phosphatase (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study.
  Measured in blood in U/L (units per liter)
Electrocardiogram (ECG) (Safety assessments) | Conducted at baseline and all monthly visits throughout the 12-month duration of the study. Additionally, the Columbia Suicide Severity Rating Scale (C-SSRS) will be administered at screening, month 6, and month 12
  Measurement of ECG QT Interval in ms (milliseconds)
Columbia Suicide Severity Rating Scale (C-SSRS) (Safety assessments) | Screening visit, month 6 and 12 months visits
  Participants will be monitored appropriately and observed for suicidal ideation and unusual behavior.

CONTACTS AND LOCATIONS:
Locations (6):
- Norway (6):
  - University Hospital of North Norway, Tromsø, Nordland
  - Akershus Hospital:, Oslo, Oslo County
  - Haugesund Hospital, Haugesund, Rogaland
  - Stavanger University Hospital, Stavanger, Rogaland
  - St. Olavs Hospital:, Trondheim, Trøndelag
  - Haraldsplass Deaconess Hospital, Bergen, Vestland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asano T, Ikegaki I, Satoh S, Suzuki Y, Shibuya M, Takayasu M, Hidaka H. Mechanism of action of a novel antivasospasm drug, HA1077. J Pharmacol Exp Ther. 1987 Jun;241(3):1033-40. PMID 3598899
- [Background] Atri A, Frolich L, Ballard C, Tariot PN, Molinuevo JL, Boneva N, Windfeld K, Raket LL, Cummings JL. Effect of Idalopirdine as Adjunct to Cholinesterase Inhibitors on Change in Cognition in Patients With Alzheimer Disease: Three Randomized Clinical Trials. JAMA. 2018 Jan 9;319(2):130-142. doi: 10.1001/jama.2017.20373. PMID 29318278
- [Background] Ballard C, Atri A, Boneva N, Cummings JL, Frolich L, Molinuevo JL, Tariot PN, Raket LL. Enrichment factors for clinical trials in mild-to-moderate Alzheimer's disease. Alzheimers Dement (N Y). 2019 May 20;5:164-174. doi: 10.1016/j.trci.2019.04.001. eCollection 2019. PMID 31193334
- [Background] Ballard C, Aarsland D, Cummings J, O'Brien J, Mills R, Molinuevo JL, Fladby T, Williams G, Doherty P, Corbett A, Sultana J. Drug repositioning and repurposing for Alzheimer disease. Nat Rev Neurol. 2020 Dec;16(12):661-673. doi: 10.1038/s41582-020-0397-4. Epub 2020 Sep 16. PMID 32939050
- [Background] Brooker H, Williams G, Hampshire A, Corbett A, Aarsland D, Cummings J, Molinuevo JL, Atri A, Ismail Z, Creese B, Fladby T, Thim-Hansen C, Wesnes K, Ballard C. FLAME: A computerized neuropsychological composite for trials in early dementia. Alzheimers Dement (Amst). 2020 Oct 14;12(1):e12098. doi: 10.1002/dad2.12098. eCollection 2020. PMID 33088895
- [Background] Corbett A, Pickett J, Burns A, Corcoran J, Dunnett SB, Edison P, Hagan JJ, Holmes C, Jones E, Katona C, Kearns I, Kehoe P, Mudher A, Passmore A, Shepherd N, Walsh F, Ballard C. Drug repositioning for Alzheimer's disease. Nat Rev Drug Discov. 2012 Nov;11(11):833-46. doi: 10.1038/nrd3869. PMID 23123941
- [Background] Couch BA, DeMarco GJ, Gourley SL, Koleske AJ. Increased dendrite branching in AbetaPP/PS1 mice and elongation of dendrite arbors by fasudil administration. J Alzheimers Dis. 2010;20(4):1003-8. doi: 10.3233/JAD-2010-091114. PMID 20413901
- [Background] Corbett A, Owen A, Hampshire A, Grahn J, Stenton R, Dajani S, Burns A, Howard R, Williams N, Williams G, Ballard C. The Effect of an Online Cognitive Training Package in Healthy Older Adults: An Online Randomized Controlled Trial. J Am Med Dir Assoc. 2015 Nov 1;16(11):990-7. doi: 10.1016/j.jamda.2015.06.014. PMID 26543007
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Elliott C, Rojo AI, Ribe E, Broadstock M, Xia W, Morin P, Semenov M, Baillie G, Cuadrado A, Al-Shawi R, Ballard CG, Simons P, Killick R. A role for APP in Wnt signalling links synapse loss with beta-amyloid production. Transl Psychiatry. 2018 Sep 20;8(1):179. doi: 10.1038/s41398-018-0231-6. PMID 30232325
- [Background] Fazekas F, Chawluk JB, Alavi A, Hurtig HI, Zimmerman RA. MR signal abnormalities at 1.5 T in Alzheimer's dementia and normal aging. AJR Am J Roentgenol. 1987 Aug;149(2):351-6. doi: 10.2214/ajr.149.2.351. PMID 3496763
- [Background] Fukumoto Y, Yamada N, Matsubara H, Mizoguchi M, Uchino K, Yao A, Kihara Y, Kawano M, Watanabe H, Takeda Y, Adachi T, Osanai S, Tanabe N, Inoue T, Kubo A, Ota Y, Fukuda K, Nakano T, Shimokawa H. Double-blind, placebo-controlled clinical trial with a rho-kinase inhibitor in pulmonary arterial hypertension. Circ J. 2013;77(10):2619-25. doi: 10.1253/circj.cj-13-0443. Epub 2013 Aug 3. PMID 23912836
- [Background] Herholz K, Salmon E, Perani D, Baron JC, Holthoff V, Frolich L, Schonknecht P, Ito K, Mielke R, Kalbe E, Zundorf G, Delbeuck X, Pelati O, Anchisi D, Fazio F, Kerrouche N, Desgranges B, Eustache F, Beuthien-Baumann B, Menzel C, Schroder J, Kato T, Arahata Y, Henze M, Heiss WD. Discrimination between Alzheimer dementia and controls by automated analysis of multicenter FDG PET. Neuroimage. 2002 Sep;17(1):302-16. doi: 10.1006/nimg.2002.1208. PMID 12482085
- [Background] Hinderling PH, Karara AH, Tao B, Pawula M, Wilding I, Lu M. Systemic availability of the active metabolite hydroxy-fasudil after administration of fasudil to different sites of the human gastrointestinal tract. J Clin Pharmacol. 2007 Jan;47(1):19-25. doi: 10.1177/0091270006293767. PMID 17192498
- [Background] Ido K, Kurogi R, Kurogi A, Nishimura K, Arimura K, Nishimura A, Ren N, Kada A, Matsuo R, Onozuka D, Hagihara A, Takagishi S, Yamagami K, Takegami M, Nohara Y, Nakashima N, Kamouchi M, Date I, Kitazono T, Iihara K; J-ASPECT Study Collaborators. Effect of treatment modality and cerebral vasospasm agent on patient outcomes after aneurysmal subarachnoid hemorrhage in the elderly aged 75 years and older. PLoS One. 2020 Apr 9;15(4):e0230953. doi: 10.1371/journal.pone.0230953. eCollection 2020. PMID 32271814
- [Background] Gillett R. Assessment of working memory performance in self-ordered selection tests. Cortex. 2007 Nov;43(8):1047-56. doi: 10.1016/s0010-9452(08)70702-0. PMID 18044665
- [Background] Grill JD, Di L, Lu PH, Lee C, Ringman J, Apostolova LG, Chow N, Kohannim O, Cummings JL, Thompson PM, Elashoff D; Alzheimer's Disease Neuroimaging Initiative. Estimating sample sizes for predementia Alzheimer's trials based on the Alzheimer's Disease Neuroimaging Initiative. Neurobiol Aging. 2013 Jan;34(1):62-72. doi: 10.1016/j.neurobiolaging.2012.03.006. Epub 2012 Apr 13. PMID 22503160
- [Background] Huentelman MJ, Stephan DA, Talboom J, Corneveaux JJ, Reiman DM, Gerber JD, Barnes CA, Alexander GE, Reiman EM, Bimonte-Nelson HA. Peripheral delivery of a ROCK inhibitor improves learning and working memory. Behav Neurosci. 2009 Feb;123(1):218-23. doi: 10.1037/a0014260. PMID 19170447
- [Background] Huntley J, Corbett A, Wesnes K, Brooker H, Stenton R, Hampshire A, Ballard C. Online assessment of risk factors for dementia and cognitive function in healthy adults. Int J Geriatr Psychiatry. 2018 Feb;33(2):e286-e293. doi: 10.1002/gps.4790. Epub 2017 Sep 27. PMID 28960500
- [Background] Ismail Z, Smith EE, Geda Y, Sultzer D, Brodaty H, Smith G, Aguera-Ortiz L, Sweet R, Miller D, Lyketsos CG; ISTAART Neuropsychiatric Symptoms Professional Interest Area. Neuropsychiatric symptoms as early manifestations of emergent dementia: Provisional diagnostic criteria for mild behavioral impairment. Alzheimers Dement. 2016 Feb;12(2):195-202. doi: 10.1016/j.jalz.2015.05.017. Epub 2015 Jun 18. PMID 26096665
- [Background] Janelidze S, Palmqvist S, Leuzy A, Stomrud E, Verberk IMW, Zetterberg H, Ashton NJ, Pesini P, Sarasa L, Allue JA, Teunissen CE, Dage JL, Blennow K, Mattsson-Carlgren N, Hansson O. Detecting amyloid positivity in early Alzheimer's disease using combinations of plasma Abeta42/Abeta40 and p-tau. Alzheimers Dement. 2022 Feb;18(2):283-293. doi: 10.1002/alz.12395. Epub 2021 Jun 20. PMID 34151519
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] Kamei S, Oishi M, Takasu T. Evaluation of fasudil hydrochloride treatment for wandering symptoms in cerebrovascular dementia with 31P-magnetic resonance spectroscopy and Xe-computed tomography. Clin Neuropharmacol. 1996 Oct;19(5):428-38. doi: 10.1097/00002826-199619050-00006. PMID 8889286
- [Background] Killick R, Ribe EM, Al-Shawi R, Malik B, Hooper C, Fernandes C, Dobson R, Nolan PM, Lourdusamy A, Furney S, Lin K, Breen G, Wroe R, To AW, Leroy K, Causevic M, Usardi A, Robinson M, Noble W, Williamson R, Lunnon K, Kellie S, Reynolds CH, Bazenet C, Hodges A, Brion JP, Stephenson J, Simons JP, Lovestone S. Clusterin regulates beta-amyloid toxicity via Dickkopf-1-driven induction of the wnt-PCP-JNK pathway. Mol Psychiatry. 2014 Jan;19(1):88-98. doi: 10.1038/mp.2012.163. Epub 2012 Nov 20. PMID 23164821
- [Background] Koster N, Knol DL, Uitdehaag BM, Scheltens P, Sikkes SA. The sensitivity to change over time of the Amsterdam IADL Questionnaire((c)). Alzheimers Dement. 2015 Oct;11(10):1231-40. doi: 10.1016/j.jalz.2014.10.006. Epub 2015 Jan 15. PMID 25598195
- [Background] Landau SM, Harvey D, Madison CM, Koeppe RA, Reiman EM, Foster NL, Weiner MW, Jagust WJ; Alzheimer's Disease Neuroimaging Initiative. Associations between cognitive, functional, and FDG-PET measures of decline in AD and MCI. Neurobiol Aging. 2011 Jul;32(7):1207-18. doi: 10.1016/j.neurobiolaging.2009.07.002. Epub 2009 Aug 5. PMID 19660834
- [Background] Morbelli S, Brugnolo A, Bossert I, Buschiazzo A, Frisoni GB, Galluzzi S, van Berckel BN, Ossenkoppele R, Perneczky R, Drzezga A, Didic M, Guedj E, Sambuceti G, Bottoni G, Arnaldi D, Picco A, De Carli F, Pagani M, Nobili F. Visual versus semi-quantitative analysis of 18F-FDG-PET in amnestic MCI: an European Alzheimer's Disease Consortium (EADC) project. J Alzheimers Dis. 2015;44(3):815-26. doi: 10.3233/JAD-142229. PMID 25362041
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Nair AB, Jacob S. A simple practice guide for dose conversion between animals and human. J Basic Clin Pharm. 2016 Mar;7(2):27-31. doi: 10.4103/0976-0105.177703. PMID 27057123
- [Background] Reijs BL, Teunissen CE, Goncharenko N, Betsou F, Blennow K, Baldeiras I, Brosseron F, Cavedo E, Fladby T, Froelich L, Gabryelewicz T, Gurvit H, Kapaki E, Koson P, Kulic L, Lehmann S, Lewczuk P, Lleo A, Maetzler W, de Mendonca A, Miller AM, Molinuevo JL, Mollenhauer B, Parnetti L, Rot U, Schneider A, Simonsen AH, Tagliavini F, Tsolaki M, Verbeek MM, Verhey FR, Zboch M, Winblad B, Scheltens P, Zetterberg H, Visser PJ. The Central Biobank and Virtual Biobank of BIOMARKAPD: A Resource for Studies on Neurodegenerative Diseases. Front Neurol. 2015 Oct 15;6:216. doi: 10.3389/fneur.2015.00216. eCollection 2015. PMID 26528237
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Schneider LS, Olin JT, Doody RS, Clark CM, Morris JC, Reisberg B, Schmitt FA, Grundman M, Thomas RG, Ferris SH. Validity and reliability of the Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S22-32. doi: 10.1097/00002093-199700112-00004. PMID 9236949
- [Background] Sellers KJ, Elliott C, Jackson J, Ghosh A, Ribe E, Rojo AI, Jarosz-Griffiths HH, Watson IA, Xia W, Semenov M, Morin P, Hooper NM, Porter R, Preston J, Al-Shawi R, Baillie G, Lovestone S, Cuadrado A, Harte M, Simons P, Srivastava DP, Killick R. Amyloid beta synaptotoxicity is Wnt-PCP dependent and blocked by fasudil. Alzheimers Dement. 2018 Mar;14(3):306-317. doi: 10.1016/j.jalz.2017.09.008. Epub 2017 Oct 19. PMID 29055813
- [Background] Smith SC, Lamping DL, Banerjee S, Harwood RH, Foley B, Smith P, Cook JC, Murray J, Prince M, Levin E, Mann A, Knapp M. Development of a new measure of health-related quality of life for people with dementia: DEMQOL. Psychol Med. 2007 May;37(5):737-46. doi: 10.1017/S0033291706009469. Epub 2006 Dec 19. PMID 17176501
- [Background] Song Y, Chen X, Wang LY, Gao W, Zhu MJ. Rho kinase inhibitor fasudil protects against beta-amyloid-induced hippocampal neurodegeneration in rats. CNS Neurosci Ther. 2013 Aug;19(8):603-10. doi: 10.1111/cns.12116. Epub 2013 May 3. PMID 23638992
- [Background] Suzuki Y, Shibuya M, Satoh S, Sugiyama H, Seto M, Takakura K. Safety and efficacy of fasudil monotherapy and fasudil-ozagrel combination therapy in patients with subarachnoid hemorrhage: sub-analysis of the post-marketing surveillance study. Neurol Med Chir (Tokyo). 2008 Jun;48(6):241-7; discussion 247-8. doi: 10.2176/nmc.48.241. PMID 18574328
- [Background] Tanaka K, Minami H, Kota M, Kuwamura K, Kohmura E. Treatment of cerebral vasospasm with intra-arterial fasudil hydrochloride. Neurosurgery. 2005 Feb;56(2):214-23; discussion 214-23. doi: 10.1227/01.neu.0000147975.24556.bc. PMID 15670369
- [Background] van Dyck CH, Swanson CJ, Aisen P, Bateman RJ, Chen C, Gee M, Kanekiyo M, Li D, Reyderman L, Cohen S, Froelich L, Katayama S, Sabbagh M, Vellas B, Watson D, Dhadda S, Irizarry M, Kramer LD, Iwatsubo T. Lecanemab in Early Alzheimer's Disease. N Engl J Med. 2023 Jan 5;388(1):9-21. doi: 10.1056/NEJMoa2212948. Epub 2022 Nov 29. PMID 36449413
- [Background] Wesnes KA, Brooker H, Ballard C, McCambridge L, Stenton R, Corbett A. Utility, reliability, sensitivity and validity of an online test system designed to monitor changes in cognitive function in clinical trials. Int J Geriatr Psychiatry. 2017 Dec;32(12):e83-e92. doi: 10.1002/gps.4659. Epub 2017 Jan 27. PMID 28128869
- [Background] Williams MM, Storandt M, Roe CM, Morris JC. Progression of Alzheimer's disease as measured by Clinical Dementia Rating Sum of Boxes scores. Alzheimers Dement. 2013 Feb;9(1 Suppl):S39-44. doi: 10.1016/j.jalz.2012.01.005. Epub 2012 Aug 1. PMID 22858530